CLINICAL TRIAL: NCT02021812
Title: Evaluation of the GORE® TAG® Thoracic Branch Endoprosthesis in the Treatment of Proximal Descending Thoracic Aortic Aneurysms
Brief Title: Feasibility Study for GORE® TAG® Thoracic Branch Endoprosthesis to Treat Proximal Descending Thoracic Aortic Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SSB 11-02
Record Dates: First submitted 2013-12-13; First posted 2013-12-27 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-08

CONDITIONS: Aortic Aneurysm, Thoracic
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Branched TAG® Device (Experimental): Treatment with the GORE® TAG® Thoracic Branch Endoprosthesis
  Interventions: Device: GORE® TAG® Thoracic Branch Endoprosthesis

INTERVENTIONS:
Device: GORE® TAG® Thoracic Branch Endoprosthesis

SUMMARY:
The purpose of this study is to assess the feasibility of the use of the GORE® TAG® Thoracic Branch Endoprosthesis to treat aneurysms involving the proximal Descending Thoracic Aorta (DTA)

DETAILED DESCRIPTION:
The GORE® TAG® Thoracic Endoprosthesis (TAG® Device) received premarket approval (PMA) for use in endovascular aneurysm repair of the descending thoracic aorta (DTA) on 23-Mar-2005 under P040043, and design changes that resulted in the conformable GORE® TAG® Thoracic Endoprosthesis (CTAG Device) received premarket approval for the treatment of aneurysms of the DTA on 23-Aug-2011 (P040043/S039). The TAG® Device and CTAG Device are intended to exclude an aneurysm from the blood circulation in patients diagnosed with DTA aneurysms. However, endovascular-only treatment options for patients with aneurysms approaching the aortic arch are limited as current stent graft technology would require coverage of the left subclavian artery (LSA) which may result in the need for a surgical revascularization procedure. This prompted the creation of the GORE® TAG® Thoracic Branch Endoprosthesis (previously known as Branched TAG® Device), which was evaluated in this study under IDE G130120 for Zone 2 aneurysms of the DTA.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of DTA aneurysm deemed to warrant surgical repair which requires proximal graft placement in Zone 2:

   1. Fusiform (≥ 55 mm), or
   2. Fusiform (>2 times native aortic diameter), or
   3. Saccular (no diameter criteria)
2. Age ≥18 years at time of informed consent signature
3. Subject is capable of complying with protocol requirements, including follow-up
4. Informed Consent Form (ICF) is signed by Subject or legal representative
5. Must have appropriate proximal aortic landing zone, defined as:

   1. Must require coverage of the left subclavian artery (LSA) origin for exclusion of the lesion
   2. Aortic inner diameters between 16-48 mm
   3. Landing zone, which must include the LSA ostium, cannot be aneurysmal, heavily calcified, or heavily thrombosed,
   4. Acceptable proximal landing zone outer curvature length for the required device
   5. Landing zone must be native aorta
6. Must have appropriate distal aortic landing zone, defined as:

   1. Outer curvature length must be ≥2cm proximal to the celiac artery
   2. Aortic inner diameters between 16-48mm (diameter should be between 16-42mm if using distal TAG® Device extension)
   3. Landing zone cannot be aneurysmal, heavily calcified, or heavily thrombosed
   4. Native aorta or previously implanted GORE® TAG® Device
7. Must have appropriate LSA landing zone, defined as:

   1. LSA length of ≥3 cm proximal to first major branch vessel if using Aortic Component with 8 mm portal diameter, or LSA length of ≥2.5 cm proximal to first major branch vessel if using Aortic Component with 12 mm portal diameter
   2. LSA inner diameters of 6-15 mm if using Aortic Component with 8 mm portal diameter, or inner diameters of 11-18 mm if using Aortic Component with 12 mm portal diameter
   3. Target branch vessel landing zone cannot be aneurysmal, heavily calcified, or heavily thrombosed

Exclusion Criteria:

1. Concomitant aneurysm/disease of the ascending aorta, aortic arch, or abdominal aorta requiring repair
2. Previous endovascular repair of the ascending aorta
3. Previous endovascular repair of the DTA with a non-Gore device
4. Surgery within 30 days of treatment
5. Infected aorta
6. Dissection of the DTA
7. Intramural hematoma of the DTA without DTA aneurysm
8. Life expectancy <2 years
9. Myocardial infarction or stroke within 6 weeks prior to treatment
10. Patient has a systemic infection and may be at increased risk of endovascular graft infection
11. Pregnant female at time of informed consent signature
12. Degenerative connective tissue disease, e.g. Marfan's or Ehler-Danlos Syndrome
13. Participation in another drug or medical device study within one year of study enrollment
14. Known history of drug abuse within one year of treatment
15. Significant thrombus or atheroma in the aortic arch
16. Tortuous or stenotic iliac and/or femoral arteries preventing introducer sheath insertion and the inability to use a conduit for vascular access
17. Planned coverage of left carotid or celiac arteries
18. Patient has known sensitivities or allergies to the device materials
19. Patient has known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment
20. Previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or known hypersensitivity to heparin
21. Diameter taper outside of the device sizing range between proximal and distal landing zones of aorta and the inability to use additional devices of different diameters to compensate for the taper
22. Mycotic aneurysm
23. Persistent refractory shock (systolic blood pressure <90 mm Hg)
24. Patient has body habitus or other medical condition which prevents adequate visualization of the aorta

    Additionally, the following exclusion criteria apply for Subjects enrolled in Stage 1:
25. Aberrant right subclavian or left vertebral arteries
26. Occluded/stenosed/hypoplastic right vertebral artery
27. Presence of a patent left internal mammary artery (LIMA) graft
28. Bilateral carotid artery disease
29. Known incomplete Circle of Willis
30. Known left vertebral artery ending in posterior inferior cerebellar artery (PICA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2022-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Dake, MD, Principal Investigator — Stanford University
Locations (6):
- United States (6):
  - Leland Stanford Junior University, Stanford, California
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - The Hitchcock Foundation (Dartmouth Hitchcock Medical Center), Lebanon, New Hampshire
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Branched TAG® Device: Treatment with the GORE® TAG® Thoracic Branch Endoprosthesis
  Branched TAG® Device
Period: Overall Study
Arm/Group | Branched TAG® Device
Started | 31
Completed | 16
Not Completed | 15
Not completed — Death | 8
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 2
Not completed — Refuse to return, COVD 19 | 2

BASELINE CHARACTERISTICS:
Arm/Group | Branched TAG® Device
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1
BMI [Mean (Standard Deviation); unit: kg/(m^2)] | 28.7 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Study Device Access
Description: Access to the aneurysm and target landing zone location is obtained via conventional vascular access and endovascular techniques.
Time Frame: During treatment procedure (day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | Branched TAG® Device
Number analyzed (Participants) | 31
Participants | 31

2. Primary Outcome: Number of Participants With Successful Study Device Deployment
Description: Absence of deployment failure will be considered a successful deployment. Deployment failure will be considered the failure of any Branched TAG® Device component (Aortic Component, Aortic Extender, or SB Component) to be released from the delivery catheter resulting in a serious adverse event (SAE) due to mechanical failure or use error.
Time Frame: During treatment procedure (day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | Branched TAG® Device
Number analyzed (Participants) | 31
Participants | 31

3. Primary Outcome: Number of Participants With Primary Procedural Side Branch Patency as Assessed by Angiography
Description: The presence of forward flow through the implanted Side Branch Component into the target branch vessel.
Time Frame: At conclusion of the treatment procedure (day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | Branched TAG® Device
Number analyzed (Participants) | 31
Participants | 31

4. Secondary Outcome: Number of Participants With 1 Month Side Branch Primary Patency Assessed by an Independent Core Lab
Time Frame: 1 Month
Measure: Count of Participants; unit: Participants
Arm/Group | Branched TAG® Device
Number analyzed (Participants) | 31
Participants | 31

5. Secondary Outcome: Number of Participants Without 1 Month Device Related Endoleaks Assessed by an Independent Core Lab
Description: Device-related endoelaks are defined as the presence of contrast within the aneurysm sac originating from the junction between any Branched TAG® Device component and the adjacent tissue (endoleak type IA or IB) OR the junction between the Aortic Component and either the SB Component or the Aortic Extender (type III endoleak).
Time Frame: 1 Month
Population: 1 participant was not assessed at 1 Month
Measure: Count of Participants; unit: Participants
Arm/Group | Branched TAG® Device
Number analyzed (Participants) | 30
Participants | 29

ADVERSE EVENTS:
Time Frame: Through 60 Months
Arm/Group | Branched TAG® Device
All-Cause Mortality (participants affected / at risk) | 8/31
Serious Adverse Events (participants affected / at risk) | 20/31
Other Adverse Events (participants affected / at risk) | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Branched TAG® Device (N=31)
Acute post hemorrhagic anemia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (2)
Cardiac arrhythmia (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 2 (2)
Heart block AV first degree (Cardiac disorders) | 1 (1)
Systolic heart failure (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Retinal vein occlusion (Eye disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Ischemic colitis (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Debility (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Unknown cause of death (General disorders) | 2 (2)
Aspiration pneumonia (Infections and infestations) | 3 (3)
Clostridium difficile infection (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (3)
Urosepsis (Infections and infestations) | 1 (1)
Anemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Hematoma traumatic (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Postoperative hypotension (Injury, poisoning and procedural complications) | 1 (1)
Procedural hemorrhage (Injury, poisoning and procedural complications) | 1 (2)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Degenerative joint disease (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower extremities weakness of (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar disc herniation (Musculoskeletal and connective tissue disorders) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CSF leakage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Paresthesia lower limb (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Device misdeployment (location) (Product Issues) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Renal disease (Renal and urinary disorders) | 1 (1)
Acute respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ascending aortic aneurysm rupture (Vascular disorders) | 1 (1)
Atherosclerotic cardiovascular disease (Vascular disorders) | 1 (1)
Brachial artery thrombosis (Vascular disorders) | 1 (1)
Hypertension worsened (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Iliac artery dissection (Vascular disorders) | 1 (1)
Leg ischemia (Vascular disorders) | 1 (1)
Peripheral ischemia (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Branched TAG® Device (N=31)
Acute post hemorrhagic anemia (Blood and lymphatic system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 5 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Macular degeneration (Eye disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Catheter site pain (General disorders) | 2 (2)
Stent-graft endoleak type IA (General disorders) | 5 (5)
Stent-graft endoleak type II (General disorders) | 5 (5)
Stent-graft endoleak type III (General disorders) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 4 (6)
Incision site hematoma (Injury, poisoning and procedural complications) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 5 (6)
Headache (Nervous system disorders) | 2 (2)
Thrombosis in device (Product Issues) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (4)
Delirium (Psychiatric disorders) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Oliguria (Renal and urinary disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Basilar atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No